CLINICAL TRIAL: NCT07294092
Title: Ketamine and Propofol NeuroImaging
Acronym: KAPNI
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Keith M Vogt (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25110029; R35GM146822 (NIH)
Record Dates: First submitted 2025-12-16; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Pain
Keywords: Propofol; Ketamine; functional MRI; electric nerve stimulation; sedation; functional connectivity
MeSH Terms: conditions — Pain | interventions — Propofol; Ketamine; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Only the ordering of drug assignments is randomized. After completing all visits, all subjects will have underwent all the same interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol, followed by propofol+ketamine (given at first visit) (Experimental): * Propofol, followed by propofol+ketamine at Visit 1
  * Ketamine, followed by ketamine+propofol at Visit 3
  * Propofol, followed by propofol+ketamine at Visit 5
  * Ketamine, followed by ketamine+propofol at Visit 7
  EEG will be done at either visits 1 and 3 or 5 and 7; fMRI will be done at the other two (non-EEG) visits.
  Interventions: Drug: Propofol; Drug: Ketamine; Device: Peripheral Nerve Stimulation
- Ketamine, followed by ketamine+propofol (given at first visit) (Experimental): * Ketamine, followed by ketamine+propofol at Visit 1
  * Propofol, followed by propofol+ketamine at Visit 3
  * Ketamine, followed by ketamine+propofol at Visit 5
  * Propofol, followed by propofol+ketamine at Visit 7
  EEG will be done at either visits 1 and 3 or 5 and 7; fMRI will be done at the other two (non-EEG) visits.
  Interventions: Drug: Propofol; Drug: Ketamine; Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Drug: Propofol — Subjects will receive an intravenous infusion of this drug, during portions of the study.
  Other Names: Diprivan
Drug: Ketamine — Subjects will receive an intravenous infusion of this drug, during portions of the study.
  Other Names: ketalar
Device: Peripheral Nerve Stimulation — Experimental acute pain stimulus will be delivered using a nerve stimulator. These painful shocks will be paired with specific experimental events.
  Other Names: electric nerve stimulation

SUMMARY:
This is a multi-visit which will collect MRI (pictures of the brain) and EEG (brain waves) data to determine changes in brain connectivity and brain activity for memory formation and pain perception while receiving the commonly-used anesthetic agents ketamine and propofol, both alone and in combination.

DETAILED DESCRIPTION:
There are four independent drug-administration sessions, visits 1, 3, 5, and 7. In all four of these sessions, both drugs are received, but in two different sequences. Two of these are EEG sessions and two are MRI sessions. Both EEG and MRI will have the same two drug orderings:

* Propofol alone, followed by ketamine and propofol together
* Ketamine alone, followed by propofol and ketamine together Assignment to propofol alone first, versus ketamine alone first will be randomized. But, all subjects will be assigned to receive both drug orderings under both EEG monitoring and MRI acquisition.

A follow-up memory testing visit will occur the day after each MRI/EEG session, on visits 2, 4, 6, and 8. No drugs are given during the next-day testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-59 years of age, who:
* have none of the specific exclusion criteria
* have a valid email address and valid phone number throughout the study
* free from any non-MRI compatible implants

Exclusion Criteria:

* are pregnant or attempting to conceive
* body mass index (BMI) > 35
* significant memory impairment or hearing loss
* sleep apnea
* chronic pain or frequently taking pain medication
* chronic medical conditions requiring treatment (hypertension, diabetes, high cholesterol)
* neurologic disease, including seizures and tremor
* psychiatric diagnoses, including anxiety, depression, panic, or PTSD
* a history of any of these medical conditions: abnormal heartbeats (cardiac conduction abnormality or arrhythmia), liver or kidney disease, or significant lung disease
* severe claustrophobia or intolerance of an MRI
* have metal implants or non-removable metal piercings
* having a history of adverse reaction to ketamine or propofol
* daily alcohol or heavy alcohol use; history of alcohol abuse
* current daily smoker
* regular or recent marijuana use (including prescribed/medical marijuana)
* illicit drug use, i.e., street drugs
* regularly taking: antiepileptics, antidepressants, anti-psychotics, antihistamines, anti-anxiety medication, stimulants, or sleep-aids

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-02 (Estimated)

PRIMARY OUTCOMES:
Explicit Memory Performance, comparing single-drug to drug-combination condition | Visits 2, 4, 6, and 8. Visits spaced at least 1 week apart, are 1 hour in length, and are 12-36 hours after the preceding visit (1, 3, 5, and 7).
  Recognition memory testing, using the Remember-Know procedure, in which subjects indicate whether they recognize previously experienced experimental items among novel items (not previously in the experiment). This allows calculation of interdependent measures of recollection & familiarity using the signal detection statistic, d'. d' is calculated as the cumulative Gaussian distribution of false positive responses subtracted from the cumulative Gaussian distribution of correctly identified previously-experienced items. d' is on a (theoretically infinite) scale of standard deviation units, with negative values representing performance worse than chance guessing and positive values representing stand deviations of performance above chance.
Pain intensity and unpleasantness ratings, comparing single-drug to drug-combination condition | Visits 1, 3, 5, and 7: immediately following each experimental condition. These visits are 3 hours in length and spaced at least 1 week apart.
  Numerical rating scale (0-10) pain score difference, comparing the single-drug condition to the steady-state dose of the drug-combination condition. Higher pain scores indicate more pain; a positive difference between pain scores during the single-drug condition minus the value during the steady-state dose of the combination-drug condition indicates pain reduction (a better outcome).

SECONDARY OUTCOMES:
MRI-based activation during memory formation, comparing the single-drug condition to the combination-drug condition | MRI visits (1 and 3, or 5 and 7), which are are 3 hours in length and spaced at least 1 week apart. Data collected at 3 timepoints in 8-minute MRI scans: at baseline, under one drug, and under both drugs.
  The Z-score is calculated by linear regression of the task timing against the MRI signal time-course (MRI data is in arbitrary units with no maximum or minimum) at each voxel (single data point in brain). Z-score of 0 indicates no task-related changes. Z-scores further from zero indicate a larger difference in brain activity, with positive values indicating decreases under the combination-drug condition, while negative Z-scores indicate increases under the combination-drug condition, compared to the single-drug condition. This outcome is reported as a number, as it is calculated using all the data across subjects combined into one statistical measure for the overall strength of difference in MRI signal change between two groups of data. Dispersion measures cannot be calculated for the summary Z-score.
MRI-based activation during painful stimulation, comparing the single-drug condition to the combination-drug condition | MRI visits (1 and 3, or 5 and 7), which are are 3 hours in length and spaced at least 1 week apart. Data collected at 3 timepoints in 8-minute MRI scans: at baseline, under one drug, and under both drugs.
  The Z-score is calculated by linear regression of the task timing against the MRI signal time-course (MRI data is in arbitrary units with no maximum or minimum) at each voxel (single data point in brain). Z-score of 0 indicates no task-related changes. Z-scores further from zero indicate a larger difference in brain activity, with positive values indicating decreases under the combination-drug condition, while negative Z-scores indicate increases under the combination-drug condition, compared to the single-drug conditions. This outcome is reported as a number, as it is calculated using all the data across subjects combined into one statistical measure for the overall strength of difference in MRI signal change between two groups of data. Dispersion measures cannot be calculated for the summary Z-score.
MRI-based changes in functional connectivity, comparing the single-drug condition to the combination-drug condition | MRI visits (1 and 3, or 5 and 7), which are are 3 hours in length and spaced at least 1 week apart. Data collected at 3 timepoints in 8-minute MRI scans: at baseline, under one drug, and under both drugs.
  Functional connectivity (FC) measures the correlation of MRI signal time-series between brain regions. Changes in FC reflect differences in brain state, in this case between single-drug and combination-drug conditions. A T-statistic of 0 indicates no change; more positive scores mean stronger connectivity in the single-drug condition, and more negative scores mean stronger connectivity with the combination-drug condition. This outcome is a number reflecting the overall magnitude of difference between two datasets, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.
EEG-based changes in functional connectivity, comparing single-drug to combination-drug condition. | EEG visits (1 and 3, or 5 and 7), which are are 3 hours in length and spaced at least 1 week apart. Data collected at 3 timepoints in 8-minute EEG scans: at baseline, under one drug, and under both drugs.
  Functional connectivity (FC) measures the correlation of MRI signal time-series between brain regions. Changes in FC reflect differences in brain state, in this case between single-drug and combination-drug conditions. A T-statistic of 0 indicates no change; more positive scores mean stronger connectivity in the single-drug condition, and more negative scores mean stronger connectivity with the combination-drug condition. This outcome is a number reflecting the overall magnitude of difference between two datasets, calculated in one summary statistic. Dispersion measures cannot be calculated for the T-statistic in this analysis framework.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to share:
  * age, height, weight, sex
  * survey results quantifying pain predispositions (catastrophizing, vigilance & anxiety), depression, anxiety, stress, and sleep
  * pain intensity & unpleasantness ratings
  * observer assessment of sedation ratings
  * Behavioral performance data for long-term memory
  * structural and functional MRI images
Supporting Information: Study Protocol, ICF
Time Frame: After analysis is complete and results have been published, all the above data will be shared in de-identified format, linked together by an assigned subject number.
Access Criteria: Data will be shared via a publicly-accessible online platform that allows user download at no cost.